CLINICAL TRIAL: NCT05869097
Title: Efficacy and Safety of Trifluridine/Tipiracil Plus Bevacizumab Versus Trifluridine/Tipiracil Monotherapy for Refractory Metastatic Colorectal Cancer: a Retrospective Study
Brief Title: Trifluridine/Tipiracil Plus Bevacizumab Versus Trifluridine/Tipiracil Monotherapy in Refractory Metastatic Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: Hunan Cancer Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: TDTB-colorectal cancer
Record Dates: First submitted 2023-05-11; First posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Metastatic Colorectal Adenocarcinoma
Keywords: Colorectal cancer; trifluridine/tipiracil ; bevacizumab
MeSH Terms: conditions — Colorectal Neoplasms | interventions — trifluridine tipiracil drug combination; Bevacizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TAS-102 plus BEV group: In TAS-102 plus BEV group, Patients received TAS-102 (35 mg/m²orally twice a day on days 1-5 and 8-12, every 28 days) and bevacizumab (5 mg /kg, intravenously, on days 1 and 15, every 28 days). Bevacizumab was approved to be a 30-minute intravenous infusion before TAS-102.
  Interventions: Drug: Trifluridine/Tipiracil; Drug: Bevacizumab
- TAS-102 monotherapy group: In TAS-102 monotherapy group, TAS-102 35 mg/m²orally twice a day on days 1-5 and 8-12, every 28 days were given to patients.
  Interventions: Drug: Trifluridine/Tipiracil

INTERVENTIONS:
Drug: Trifluridine/Tipiracil — TAS-102 35 mg/m²orally twice a day on days 1-5 and 8-12, every 28 days
  Other Names: TAS-102; Lonsurf; S 95005
Drug: Bevacizumab — Bevacizumab 5 mg /kg, intravenously on days 1,15,every 28 days
  Other Names: Avastin
  Groups: TAS-102 plus BEV group

SUMMARY:
This study is a retrospective study to compare the efficacy and safety between trifluridine/tipiracil (TAS-102) plus bevacizumab (BEV) with TAS-102 monotherapy in refractory metastatic colorectal cancer (mCRC) from November 2020 to October 2022 at the Hunan Cancer Hospital.

DETAILED DESCRIPTION:
Our retrospective analysis was conducted to explore the efficacy and safety of patients treated with at least 1 cycle of TAS-102 with or without BEV in patients suffering refractory mCRC from November 2020 to October 2022 at the Hunan Cancer Hospital. Data from the electronic medical records were the sources. In TAS-102 monotherapy group, TAS-102 35 mg/m²orally twice a day on days 1-5 and 8-12, every 28 days were given to patients, while on days 1 and 15, every 28 days, patients received bevacizumab (5 mg /kg, intravenously) in TAS-102 plus BEV group. The median OS (mOS) was the primary end point.while mPFS, the ORR, the disease control rate(DCR) and the incidence of treatment-related adverse events (TRAEs) were the secondary end points.

ELIGIBILITY:
Inclusion Criteria:

* 1.Has histologically confirmed unresectable adenocarcinoma of the colon or rectum (all other histological types are excluded).

  2. Have progressed from at least 2 lines of standard treatment,including fluoropyrimidines, irinotecan, oxaliplatin, with or without targeted drugs, like bevacizumab and cetuximab (only for RAS wild-type). Fruquintinib or regorafenib was permitted but not required for inclusion.

  3.Has measurable or non-measurable disease as defined by RECIST version 1.1 4.Is able to swallow oral tablets. 5.Estimated life expectancy ≥12 weeks. 6.Eastern Cooperative Oncology Group performance status (ECOG PS) 0 or 1 7. Has adequate organ function.

Exclusion Criteria:

* 1.Pregnancy, lactating female or possibility of becoming pregnant during the study.

  2.Has not recovered from clinically relevant non-hematologic CTCAE grade ≥ 3 toxicity of previous anticancer therapy (excluding alopecia, and skin pigmentation).

  3.Has symptomatic central nervous system metastases that are neurologically unstable or requiring increasing doses of steroids to control CNS disease.

  4.Has severe or uncontrolled active acute or chronic infection. 5.Known carriers of HIV antibodies. 6.Confirmed uncontrolled arterial hypertension or uncontrolled or symptomatic arrhythmia.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population were the patients treated with at least 1 cycle of TAS-102 with or without BEV in patients suffering refractory mCRC from November 2020 to October 2022 at the Hunan Cancer Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) | Approximately 12 months
  Overall survival defined as the observed time elapsed between the date of commencement of treatment and the date of death due to any cause

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Approximately 12 months
  Progression-free survival defined as the time elapsed between the date of commencement of treatment and the date of radiologic tumour progression according to RECIST version 1.1 by investigator's judgement or death from any cause, whichever comes first.
Overall response rate (ORR) | Approximately 12 months
  Overall response rate (ORR) was regarded as the proportion of complete responses (CRs) and partial responses (PRs) according to RECIST version 1.1 criteria and using investigator's tumor assessment
Disease control rate (DCR) | Approximately 12 months
  Disease control rate has been defined as the addition of (CR + PR) rate and also stable disease (SD) rate
Treatment-Related Adverse Events (TRAE) | Approximately 12 months
  Treatment-Related Adverse Events (TRAE) as assessed by CTCAE v5.0, including serious adverse events (SAEs)

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan Cancer hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for principal investigator or correspondence author]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: please contact the principal investigator of this study or correspondence author.